CLINICAL TRIAL: NCT06446479
Title: Effects of THC on Alcohol Consumption and Neural Correlates of Reward
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 22-1314
Record Dates: First submitted 2024-02-13; First posted 2024-06-06 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Cannabis Use Disorder
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo first, Dronabinol second (Experimental): This arm will receive placebo on the first visit, and dronabinol on the second visit
  Interventions: Drug: Dronabinol Pill; Drug: Placebo
- Dronabinol first, Placebo second (Experimental): This arm will receive dronabinol on the first visit, and placebo on the second visit.
  Interventions: Drug: Dronabinol Pill; Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol Pill — Dronabinol 20 mg
Drug: Placebo — placebo

SUMMARY:
Alcohol and cannabis are often used together such that their effects overlap, but little is known about the neural mechanisms that underlie simultaneous use. High doses of THC have not been well-studied in the laboratory, and it is unclear how high doses of THC may impact alcohol consumption patterns. The proposed study will explore the effects of oral THC (20mg dronabinol) vs. placebo on neural reward, alcohol self-administration and naturalistic co-use patterns.

DETAILED DESCRIPTION:
Participants will undergo a screening assessment, baseline session and two laboratory visits. The laboratory visits will involve an MRI scan and the opportunity to consume alcohol in our BAR lab. Prior to the MRI, participants will consume, a placebo (0mg) or high (20mg) dose of oral THC (dronabinol). Visits will be separated by 7 to 14 days. Dronabinol is an FDA-approved product that will be dispensed by our on-campus pharmacy

ELIGIBILITY:
Inclusion Criteria:

* Drink alcohol
* Use cannabis
* Contact site for additional details

Exclusion Criteria:

* MRI contraindications (implanted metal, weight > 315 lb, etc.).
* Contact site for additional details

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol cue-elicited brain activation (fMRI) between medication periods | 1 hour after administration of a single dose of study medication at 7 days, 14 days.
  Alcohol cue reactivity task BOLD signal to alcohol cues, relative to neutral beverage cues
Change in cannabis cue-elicited brain activation (fMRI) between medication periods | 1 hour after administration of a single dose of study medication at 7 days, 14 days.
  Cannabis cue reactivity task BOLD signal to cannabis cues, relative to neutral cues
Alcohol self-administration | 3-4 hours after administration of a single dose of study medication at 7 days, 14 days.
  Number of drinks self-administered
Self-reported alcoholic drinks consumed | one report per day for the 14 days after the final laboratory visit on day 14.
  # of drinks consumed per day
Self-reported cannabis use | One report per day for the 14 days after the final laboratory visit on day 14
  Amount of cannabis consumed per day
Self-reported cannabis and alcohol co-use | One report per day for the 14 days after the final laboratory visit on day 14.
  Number of days in which cannabis and alcohol were both used

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States